CLINICAL TRIAL: NCT05282849
Title: Ultrasound Guided Quadratus Lumborum Block Versus Fascia Iliaca Block in Pediatric Patients Undergoing Developmental Dysplasia of Hip Surgical Repair. A Randomized Comparative Study
Brief Title: Ultrasound Quadratus Lumborum Block Vs Fascia Iliaca Block in Pediatrics Undergoing Hip Surgery .
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Mohamed Abd El Moneim Soaida, MD, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMS2022-1
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Developmental Dysplasia of the Hip
Keywords: ultrasound; quadratus lumborum; fascia iliaca
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group F: ultrasound guided fascia iliaca block group (Active Comparator)
  Interventions: Procedure: ultrasound guided fascia iliaca block
- Group Q: ultrasound guided quadratus lumborum block group (Active Comparator)
  Interventions: Procedure: ultrasound guided quadratus lumborum block

INTERVENTIONS:
Procedure: ultrasound guided fascia iliaca block — ultrasound guided fascia iliaca block anesthetizes variable combinations of the femoral nerve , lateral femoral cutaneous nerve , and obturator nerve, and is effective for many painful hip surgeries making it potentially useful for analgesia following Developmental Dysplasia of Hip (DDH) surgery.
  Arms: Group F: ultrasound guided fascia iliaca block group
Procedure: ultrasound guided quadratus lumborum block — ultrasound-guided quadratus lumborum (QL) block provides perioperative somatic, even visceral analgesia for patients including pediatrics, undergoing abdominal or hip surgery. The local anesthetic injected adjacently into the quadrates lumborum muscle spreads in a medial and cranial direction under the crura and arcuate ligaments of the diaphragm, then into the thoracic paravertebral space anesthetizing the hip region
  Arms: Group Q: ultrasound guided quadratus lumborum block group

SUMMARY:
Comparison between ultrasound guided transmuscular QL block and Fascia iliaca block in pediatric patients undergoing DDH surgery regarding the quality of pain control in the perioperative period..

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-12 years
* Of both sexes
* American society of anesthesiologist (ASA) physical status classification class I
* Undergoing general anaesthesia for DDH surgery

Exclusion Criteria:

* Parents' refusal of regional block
* Duration of surgery over 120 min.
* History of allergy to local anesthetics
* Bleeding disorders (INR >1.4, Platelet count< 75000)

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Total 12 hours postoperative opioid consumption | from the time of transfer of the patient to the pacu at one hour intervals for 12 hours
  amount of morphine consumed as rescue analgesia in first 12 hours

SECONDARY OUTCOMES:
Postoperative pain using Face, Legs, Activity, Cry, Consolability scale (FLACC ) pain rating scale | from the time of transfer to the PACU, every hour for the first 24 hours postoperative]
  pain score of paitients in the post operative period
Side effects | from the time of transfer to the PACU, for the first 24 hours postoperative
  respiratory depression and postoperative nausea and vomiting
Total 24 hours postoperative opioid consumption | from the time of transfer of the patient to the pacu at one hour intervals for 24hours
  amount of morphine consumed as rescue analgesia in first 24hours

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided